CLINICAL TRIAL: NCT00933621
Title: Intracoronary Injection of Autologous Bone Marrow Cells in Patients With Chronic Heart Failure: Five Years Follow up
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Alex Blatt, Assaf Harofeh MC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-03
Record Dates: First submitted 2009-06-30; First posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Ischemic Symptomatic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Bone Marrow infusion (Experimental): Percutaneous intracoronary autologous bone marrow infusion
  Interventions: Procedure: Autologous bone marrow intracoronary infusion

INTERVENTIONS:
Procedure: Autologous bone marrow intracoronary infusion — Percutaneous intracoronary mononuclear bone marrow cell infusion
  Other Names: Intracoronary mononuclear bone marrow cell infusion

SUMMARY:
The study aim is to evaluate the long term outcome of intra-coronary autologous bone marrow (BM) transplantation in patients with severe ischemic cardiomyopathy without the option for revascularization.

DETAILED DESCRIPTION:
Several studies have demonstrated the short term safety, feasibility and efficacy of cell transplantation in patients with advanced heart failure. There are no data about the long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of hibernation and/or ischemia in at least 2 different myocardial segments underwent coronary angiography

Exclusion Criteria:

* Idiopathic or non-ischemic cardiomyopathy
* Other etiology for heart failure, history of past or current disease involving the bone marrow
* Patients on dialysis
* Positive serologic test for HIV, hepatitis B or C or any neoplastic or terminal disease

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-04; Primary Completion 2003-05 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Procedure success | 9 months

SECONDARY OUTCOMES:
Functional class improvement | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex Blatt, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Assaf Harofeh, Ẕerifin, Israel

REFERENCES:
- [Background] Abdel-Latif A, Bolli R, Tleyjeh IM, et al. Adult bone marrow-derived cells for cardiac repair. Arch Intern Med. 2007;167:989-997. 12. Murry CE, Reinecke H and Pabon LM. Regeneration Gaps: Observation on stem cells and cardiac repair. J Am Coll Cardiol. 2006;47:1777-1785.